CLINICAL TRIAL: NCT05080335
Title: Transgender and Gender-expansive Youth: Randomized Controlled Trial of a Healthcare Didactic Enhanced by Simulated Patient Video Clips
Brief Title: Transgender Health: an Educational RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2000028980_c
Record Dates: First submitted 2021-09-22; First posted 2021-10-15 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Transgender; Health Attitude

STUDY DESIGN:
Intervention Model Description: RCT of three different education / training approaches
Who Masked: Participant, Investigator
Masking Description: Participants will not be aware of which of the four arms they will be assigned to
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- TRANS-gender female instructor, with videos (TV) (Active Comparator): Didactic materials use embedded WITH short videos of transgender youth; lesson led by a TRANS-gender woman with extensive experience as an educator on transgender health
  Interventions: Other: Short videos
- CIS-gender female instructor, with videos (CV) (Active Comparator): Didactic materials use embedded WITH short videos of transgender youth; lesson led by a CIS-gender woman with extensive experience as an educator on transgender health
  Interventions: Other: Short videos
- CIS-gender female, with NO videos (CN) (Active Comparator): Didactic materials do NOT use short videos of transgender youth [until AFTER completion of the POST outcome measures]; lesson is led by a CIS-gender woman with extensive experience as an educator on transgender health
  Interventions: Other: Short videos
- No intervention control (No Intervention): Subjects randomized to this arm will complete the baseline assessment and the post assessment thirty days later, but just *before* receiving the intervention (TV).

INTERVENTIONS:
Other: Short videos — As an educational RCT, the didactic content will be the same across the four arms, but its deliver will vary by:
  1. TRANS- vs CIS-gender female instructors
  2. With or without short videos of transgender youth embedded into the didactic [TV or CV]; for the group with no embedded videos [NV], the same videos will be shown AFTER completion of the post measures)
  3. No-intervention control, in which TV will be delivered *after* collection of pre/post measures.
  Arms: CIS-gender female instructor, with videos (CV); CIS-gender female, with NO videos (CN); TRANS-gender female instructor, with videos (TV)

SUMMARY:
The investigators will conduct a randomized controlled trial (RCT) comparing two different educational approaches on the healthcare of transgender and gender expansive (TGE) youth. Finding best practices to educate healthcare providers and the community at large stand to make an impact on the mental health of TGE youth by helping them feel more welcome and better understood by the communities in which they live.

The study aims are to evaluate two educational interventions: 1) The inclusion of a video clip component of two TGE youth (Video [V] vs No video [N]) into a one-hour didactic; and 2) The delivery of the same didactic content by a cis- [C] vs a trans-gender [TG] woman.

DETAILED DESCRIPTION:
This will be a randomized control trial (RCT) of equal allotment to one of four parallel didactic conditions. The investigators will randomly assign participants to one of three teaching conditions: 1) Trans Video [TV]; 2) Cis Video [CV]; and 3) Cis No video [CN]. Participants will complete a baseline assessment (PRE) before the start of the same didactic content, but delivered in the three different ways described above. This design will help the investigators make comparisons across video use (yes/no), about type of presenter (trans/cis), and about the interaction of the two approaches. For the 'no video' condition (CN), the didactic will not include the videos until after completion of the POST assessment.

The study design will ensure that all participants will receive the exact same didactic content during whichever session they attend. All participants will then receive a follow up questionnaire two weeks later (2WK POST) to assess content retention.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Living in the US
* Ages GE 18

Exclusion Criteria:

* None

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Change in T-KAB TOTAL score (TOT) | Before / after viewing videos (within 60 minutes), and after 30 days.
  The T-KAB (Clark and Hughto, 2020) is a 22-item, 3-factor measure representing: acceptance of the gender spectrum (ACC), social tolerance (ST), and comfort and contact (CC) related to transgender people. The total score (TOT) is the sum of it three sub-scales.
  The adjusted T-KAB It is scored on a 6-point Likert scale (instead of the 4-point original) ranging from 1 ("Strongly disagree") to 4 ("Strongly agree"). An even-number scale was utilized to ensure that participants choose either agreement or disagreement, and thus, a neutral option was not included in the scale.
  This results in an item-level score ranging from 1 to 6, and an overall TOT range from 22 to 132, with higher numbers representing better outcomes.
  We changed the wording and reverse-scoring of 6 items, which due to double-negative wording, proved confusing in pilot testing. This resulted in 9/22 reverse-scored items (R), from the original scale with 15/22 R's.

SECONDARY OUTCOMES:
Change in T-KAB ACCEPTANCE sub-scale (ACC) | Before / after viewing videos (within 60 minutes), and after 30 days.
  The T-KAB ACCEPTANCE sub-scale (ACC) is an 8-item measure representing acceptance of the gender spectrum
  The adjusted ACC is scored on a 6-point Likert scale ranging from 1 ("Strongly disagree") to 6 ("Strongly agree"). This adjustment resulted in an item-level score ranging from 1 to 6, and an overall TOT ranging from 8 to 48, with higher numbers representing better acceptance of the gender spectrum.
  Of note, all six items changed from double negative wording were part of the ACC sub-scale. As one example, we changed ACC item 1 from:
  A person with a vagina cannot can be a man. (R)
  to:
  A person with a vagina can can be a man.
Change in T-KAB SOCIAL TOLERANCE sub-scale (ST) | Before / after viewing videos (within 60 minutes), and after 30 days.
  The T-KAB SOCIAL TOLERANCE sub-scale (ST) is a 7-item measure representing social tolerance (ST) related to transgender people.
  The adjusted ST is scored on a 6-point Likert scale ranging from 1 ("Strongly disagree") to 6 ("Strongly agree"). This adjustment resulted in an item-level score ranging from 1 to 6, and an overall TOT ranging from 7 to 42, with higher numbers representing better social tolerance related to transgender individuals.
Change in T-KAB COMFORT AND CONTACT sub-scale (CC) | Before / after viewing videos (within 60 minutes), and after 30 days.
  The T-KAB COMFORT AND CONTACT sub-scale (CC) is a 7-item measure representing social tolerance (ST) related to transgender people.
  The adjusted ST is scored on a 6-point Likert scale ranging from 1 ("Strongly disagree") to 6 ("Strongly agree"). This adjustment resulted in an item-level score ranging from 1 to 6, and an overall TOT ranging from 7 to 42, with higher numbers representing better comfort and contact related to transgender individuals.
Change in SOCIAL comfort level (SOC) | Before / after viewing videos (within 60 minutes), and after 30 days.
  This item uses a slider ranging continuously from 0 ("Very uncomfortable") to 100 ("Very comfortable") in response to the question "How comfortable would you be interacting SOCIALLY with transgender individuals?") Higher numbers indicate higher comfort level.
Change in PROFESSIONAL comfort level (PROF) | Before / after viewing videos (within 60 minutes), and after 30 days.
  This item uses a slider ranging continuously from 0 ("Very uncomfortable") to 100 ("Very comfortable") in response to the question "How comfortable would you be interacting in a PROFESSIONAL or EDUCATIONAL setting with transgender individuals?") Higher numbers indicate higher comfort level.
Change in FAMILIAL comfort level (FAM) | Before / after viewing videos (within 60 minutes), and after 30 days.
  This item uses a slider ranging continuously from 0 ("Very uncomfortable") to 100 ("Very comfortable") in response to the question "How comfortable would you be interacting with a transgender individual in your FAMILY ") Higher numbers indicate higher comfort level.

OTHER OUTCOMES:
SOCIAL TOLERANCE Item 1 (SOC_01) | Before / after viewing videos (within 60 minutes), and after 30 days.
  Response to the stem:
  Transgender people should have the opportunity to undergo operations to change their anatomy.
  Scoring on a 6-point Likert scale ranging from 1 ("Strongly disagree") to 6 ("Strongly agree"), resulting in a score ranging from 1 to 6 with higher numbers representing better comfort and contact related to transgender individuals.
SOCIAL TOLERANCE Item 2 (SOC_02) | Before / after viewing videos (within 60 minutes), and after 30 days.
  Response to the stem:
  Transgender people should be accepted completely into our society.
  Scoring on a 6-point Likert scale ranging from 1 ("Strongly disagree") to 6 ("Strongly agree"), resulting in a score ranging from 1 to 6 with higher numbers representing better comfort and contact related to transgender individuals.
SOCIAL TOLERANCE Item 3 (SOC_03) | Before / after viewing videos (within 60 minutes), and after 30 days.
  Response to the stem:
  Transgender people should have the opportunity to change their name.
  Scoring on a 6-point Likert scale ranging from 1 ("Strongly disagree") to 6 ("Strongly agree"), resulting in a score ranging from 1 to 6 with higher numbers representing better comfort and contact related to transgender individuals.
SOCIAL TOLERANCE Item 4 (SOC_04) | Before / after viewing videos (within 60 minutes), and after 30 days.
  Response to the stem:
  Organizations that promote transgender rights are necessary.
  Scoring on a 6-point Likert scale ranging from 1 ("Strongly disagree") to 6 ("Strongly agree"), resulting in a score ranging from 1 to 6 with higher numbers representing better comfort and contact related to transgender individuals.
SOCIAL TOLERANCE Item 5 (SOC_05) | Before / after viewing videos (within 60 minutes), and after 30 days.
  Response to the stem:
  It should be illegal for people to have their genitalia surgically altered. (R)
  Scoring on a 6-point Likert REVERSED scale ranging from 1 ("Strongly agree") to 6 ("Strongly disagree"), resulting in a score ranging from 1 to 6 with higher numbers representing better comfort and contact related to transgender individuals.
SOCIAL TOLERANCE Item 6 (SOC_06) | Before / after viewing videos (within 60 minutes), and after 30 days.
  Response to the stem:
  Being transgender is a sin. (R)
  Scoring on a 6-point Likert REVERSED scale ranging from 1 ("Strongly agree") to 6 ("Strongly disagree"), resulting in a score ranging from 1 to 6 with higher numbers representing better comfort and contact related to transgender individuals.
SOCIAL TOLERANCE Item 7 (SOC_07) | Before / after viewing videos (within 60 minutes), and after 30 days.
  Response to the stem:
  Transgender people are a worthwhile part of our society.
  Scoring on a 6-point Likert scale ranging from 1 ("Strongly disagree") to 6 ("Strongly agree"), resulting in a score ranging from 1 to 6 with higher numbers representing better comfort and contact related to transgender individuals.
COMFORT and CONTACT Item 8 (CC_08) | Before / after viewing videos (within 60 minutes), and after 30 days.
  Response to the stem:
  I avoid interacting with people whose gender is unclear to me. (R)
  Scoring on a 6-point Likert REVERSED scale ranging from 1 ("Strongly agree") to 6 ("Strongly disagree"), resulting in a score ranging from 1 to 6 with higher numbers representing better comfort and contact related to transgender individuals.
COMFORT and CONTACT Item 9 (CC_09) | Before / after viewing videos (within 60 minutes), and after 30 days.
  Response to the stem:
  People with both breasts and a penis make me uncomfortable. (R)
  Scoring on a 6-point Likert REVERSED scale ranging from 1 ("Strongly agree") to 6 ("Strongly disagree"), resulting in a score ranging from 1 to 6 with higher numbers representing better comfort and contact related to transgender individuals.
COMFORT and CONTACT Item 10 (CC_10) | Before / after viewing videos (within 60 minutes), and after 30 days.
  Response to the stem:
  When I meet someone, it is important for me to be able to identify them as a man or a woman. (R)
  Scoring on a 6-point Likert REVERSED scale ranging from 1 ("Strongly agree") to 6 ("Strongly disagree"), resulting in a score ranging from 1 to 6 with higher numbers representing better comfort and contact related to transgender individuals.
COMFORT and CONTACT Item 11 (CC_11) | Before / after viewing videos (within 60 minutes), and after 30 days.
  Response to the stem:
  I feel uncomfortable when I cannot tell if someone is a man or a woman. (R)
  Scoring on a 6-point Likert REVERSED scale ranging from 1 ("Strongly agree") to 6 ("Strongly disagree"), resulting in a score ranging from 1 to 6 with higher numbers representing better comfort and contact related to transgender individuals.
COMFORT and CONTACT Item 12 (CC_12) | Before / after viewing videos (within 60 minutes), and after 30 days.
  Response to the stem:
  I would feel uncomfortable if a close family member were dating a transgender person. (R)
  Scoring on a 6-point Likert REVERSED scale ranging from 1 ("Strongly agree") to 6 ("Strongly disagree"), resulting in a score ranging from 1 to 6 with higher numbers representing better comfort and contact related to transgender individuals.
COMFORT and CONTACT Item 13 (CC_13) | Before / after viewing videos (within 60 minutes), and after 30 days.
  Response to the stem:
  I would feel comfortable if I learned a friend is transgender.
  Scoring on a 6-point Likert scale ranging from 1 ("Strongly disagree") to 6 ("Strongly agree"), resulting in a score ranging from 1 to 6 with higher numbers representing better comfort and contact related to transgender individuals.
COMFORT and CONTACT Item 14 (CC_14) | Before / after viewing videos (within 60 minutes), and after 30 days.
  Response to the stem:
  I would feel comfortable if I learned my neighbor is transgender.
  Scoring on a 6-point Likert scale ranging from 1 ("Strongly disagree") to 6 ("Strongly agree"), resulting in a score ranging from 1 to 6 with higher numbers representing better comfort and contact related to transgender individuals.
ACCEPTANCE Item 15 (ACC_15) | Before / after viewing videos (within 60 minutes), and after 30 days.
  Response to the stem:
  A person with a vagina can be a man.
  Scoring on a 6-point Likert scale ranging from 1 ("Strongly disagree") to 6 ("Strongly agree"), resulting in a score ranging from 1 to 6 with higher numbers representing better acceptance of the gender spectrum.
ACCEPTANCE Item 16 (ACC_16) | Before / after viewing videos (within 60 minutes), and after 30 days.
  Response to the stem:
  A person with a penis can be a woman.
  Scoring on a 6-point Likert scale ranging from 1 ("Strongly disagree") to 6 ("Strongly agree"), resulting in a score ranging from 1 to 6 with higher numbers representing better acceptance of the gender spectrum.
ACCEPTANCE Item 17 (ACC_17) | Before / after viewing videos (within 60 minutes), and after 30 days.
  Response to the stem:
  Female-to-male transgender people are real men.
  Scoring on a 6-point Likert scale ranging from 1 ("Strongly disagree") to 6 ("Strongly agree"), resulting in a score ranging from 1 to 6 with higher numbers representing better acceptance of the gender spectrum.
ACCEPTANCE Item 18 (ACC_18) | Before / after viewing videos (within 60 minutes), and after 30 days.
  Response to the stem:
  Male-to-female transgender people are real women.
  Scoring on a 6-point Likert scale ranging from 1 ("Strongly disagree") to 6 ("Strongly agree"), resulting in a score ranging from 1 to 6 with higher numbers representing better acceptance of the gender spectrum.
ACCEPTANCE Item 19 (ACC_19) | Before / after viewing videos (within 60 minutes), and after 30 days.
  Response to the stem:
  A person transitioning from female to male should be able to use a men's bathroom.
  Scoring on a 6-point Likert scale ranging from 1 ("Strongly disagree") to 6 ("Strongly agree"), resulting in a score ranging from 1 to 6 with higher numbers representing better acceptance of the gender spectrum.
ACCEPTANCE Item 20 (ACC_20) | Before / after viewing videos (within 60 minutes), and after 30 days.
  Response to the stem:
  There are only two genders: male and female.
  Scoring on a 6-point Likert REVERSED scale ranging from 1 ("Strongly agree") to 6 ("Strongly disagree"), resulting in a score ranging from 1 to 6 with higher numbers representing better comfort and contact related to transgender individuals.
ACCEPTANCE Item 21 (ACC_21) | Before / after viewing videos (within 60 minutes), and after 30 days.
  Response to the stem:
  Sex and gender are the same thing.
  Scoring on a 6-point Likert REVERSED scale ranging from 1 ("Strongly agree") to 6 ("Strongly disagree"), resulting in a score ranging from 1 to 6 with higher numbers representing better comfort and contact related to transgender individuals.
ACCEPTANCE Item 22 (ACC_22) | Before / after viewing videos (within 60 minutes), and after 30 days.
  Response to the stem:
  A person transitioning from male to female should be able to use a women's bathroom.
  Scoring on a 6-point Likert scale ranging from 1 ("Strongly disagree") to 6 ("Strongly agree"), resulting in a score ranging from 1 to 6 with higher numbers representing better acceptance of the gender spectrum.

CONTACTS AND LOCATIONS:
Overall Officials: Andres Martin, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Yale Child Center, New Haven, Connecticut
  - Yale Child Study Center, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clark, K.A., Hughto, J.M. Development and Psychometric Evaluation of the Transgender Knowledge, Attitudes, and Beliefs (T-KAB) Scale. Sex Res Soc Policy 17, 353-363 (2020). — https://doi.org/10.1007/s13178-019-00399-9